CLINICAL TRIAL: NCT01821222
Title: Mobile Phones as a Health Communication Tool to Improve Maternal and Neonatal Health in Zanzibar
Brief Title: Wired Mothers - Use of Mobile Phones to Improve Maternal and Neonatal Health in Zanzibar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Ministry of Health and Social Welfare, Zanzibar (Other Government); Danish International Development Cooperation (Unknown)
Responsible Party: Principal Investigator, Stine Lund, MD, PhD fellow, MD, PhD fellow, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-086KU
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Pregnancy; Maternal Health; Newborn Death; Health Behavior; mHealth
Keywords: Maternal health; Neonatal health; mHealth; Mobile phones; Access to health services; Health behavior
MeSH Terms: conditions — Perinatal Death; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wired mothers intervention (Experimental): The wired mothers' intervention consisted of two components: an automated short messaging service (SMS) system providing wired mothers with unidirectional text messaging and a mobile phone voucher system providing the possibility of direct two-way communication between wired mothers and their primary health care providers. While only women with registered phone numbers received text messages, all women in the intervention group were given mobile phone vouchers to contact their local primary health care provider.
  Interventions: Device: Wired mothers
- Control (No Intervention): The control group received standard care

INTERVENTIONS:
Device: Wired mothers — The wired mothers SMS component provided health education and appointment reminders to encourage attendance at routine antenatal care, skilled delivery attendance and postnatal care. A specially-designed software automatically generated and sent text messages throughout the pregnancy until six weeks after delivery. The frequency and content of the messages varied according to the women's gestational age.
  Mobile phone vouchers allowed all wired mothers to communicate directly with primary health care providers. Primary health care facilities randomised for intervention and hospitals were provided with a mobile phone with sufficient credit, while wired mothers were given a phone voucher with modest credit and a card with the phone number of her local primary health care provider.
  Arms: Wired mothers intervention

SUMMARY:
Reducing maternal and newborn mortality remains a global challenge. Because obstetric complications cannot be predicted, skilled attendance at the time of delivery and access to emergency obstetric care remain the most effective strategies to reduce mortality. Antenatal care has the potential to reduce maternal morbidity and improve newborns survival but this benefit may not be realized in sub-Saharan Africa where the attendance and quality of care is declining. There is a rapidly expanding number of mobile phone users in developing countries and due to the potential to strengthen health system the use of mobile phones is health care is emerging. The investigators assessed a mobile phone intervention named "wired mothers" aimed to improve maternal and newborn health.

The hypothesis of the study was that the wired mothers mobile phone intervention would increase attendance to essential reproductive health services such as antenatal care and skilled delivery attendance and reduce severe adverse pregnancy outcomes for women and newborn.

The objective of the study was to examine the effect of the wired mothers intervention on antenatal care, skilled delivery attendance, access to emergency obstetric care and perinatal mortality.

The study was a pragmatic cluster randomized controlled trial with the primary health care facility as the unit of randomization. The study took place in 2009-2010 on the island of Unguja in Zanzibar. 2550 pregnant women who attended antenatal care at one of 24 selected facilities were included at their first visit and followed until 42 days after delivery. Facilities were allocated by simple randomization to either mobile phone intervention (n=12) or standard care (n=12). The intervention consisted of a SMS and mobile phone voucher component.

The perspectives of the study are that mobile phones may contribute to saving the lives of women and their newborns and achievement of MDGs 4 and 5. Evidence is needed to guide maternal and child health policy makers in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending antenatal care at one of 24 selected primary healthcare facilities

Exclusion Criteria:

* Missing end-of-study questionnaire

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2550 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Skilled delivery attendance | From inclusion to 42 days after delivery. Asssessed at delivery and confirmed 42 days after delivery
  We used the WHO definition, whereby skilled delivery attendants are midwifes, doctors or nurses who have been educated and trained in the skills needed to manage pregnancies, childbirth and complications in women and newborns. We also included home deliveries assisted by skilled birth attendants, although international consensus has not been reached on this issue.

SECONDARY OUTCOMES:
Perinatal mortality | From inclusion of the pregnant women until 7 days after delivery. Assessed at delivery and 7 days after delivery
  Calculated as a composite of stillbirths and early neonatal deaths
Antenatal care attendance | From inclusion of the pregnant women until delivery

OTHER OUTCOMES:
Anti tetanus vaccination | From inclusion of the pregnant women until delivery
Preventive malaria treatment | From inclusion of the pregnant women until delivery
Antepartum and intrapartum referrals | From inclusion of the pregnant women until postpartum period
Number of calls between women and midwifes | From inclusion of the pregnant women until 42 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Stine Lund, MD, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- 24 Primary Healthcare Facilities on the island on Unguja, Zanzibar, Tanzania

REFERENCES:
- [Result] Lund S, Hemed M, Nielsen BB, Said A, Said K, Makungu MH, Rasch V. Mobile phones as a health communication tool to improve skilled attendance at delivery in Zanzibar: a cluster-randomised controlled trial. BJOG. 2012 Sep;119(10):1256-64. doi: 10.1111/j.1471-0528.2012.03413.x. Epub 2012 Jul 17. PMID 22805598
- [Derived] Lund S, Rasch V, Hemed M, Boas IM, Said A, Said K, Makundu MH, Nielsen BB. Mobile phone intervention reduces perinatal mortality in zanzibar: secondary outcomes of a cluster randomized controlled trial. JMIR Mhealth Uhealth. 2014 Mar 26;2(1):e15. doi: 10.2196/mhealth.2941. PMID 25098184
- [Derived] Lund S, Nielsen BB, Hemed M, Boas IM, Said A, Said K, Makungu MH, Rasch V. Mobile phones improve antenatal care attendance in Zanzibar: a cluster randomized controlled trial. BMC Pregnancy Childbirth. 2014 Jan 17;14:29. doi: 10.1186/1471-2393-14-29. PMID 24438517